CLINICAL TRIAL: NCT03394651
Title: The Current Status and Progression of Symptoms and Comorbidities Among Male Lower Urinary Tract Symptoms Patients in China: a Multicenter Study From Prostatic Obstruction Investigation Team (POInT)
Brief Title: Prostatic Obstruction Investigation Team Multicenter Study
Acronym: POInT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: Beijing Hospital (Other Government); Zhongda Hospital (Other); RenJi Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); The Second Hospital of Nanjing Medical University (Other); Shanghai Changzheng Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); First Affiliated Hospital of Suzhou Medical College (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Zhujiang Hospital (Other); Zhejiang University (Other); Shanghai Zhongshan Hospital (Other); Xinqiao Hospital of Chongqing (Other); Zhejiang Provincial People's Hospital (Other); Huashan Hospital (Other); Southwest Hospital, China (Other); First Affiliated Hospital of Fujian Medical University (Other); The First Affiliated Hospital of Beijing University (Unknown); Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other); Tianjin Medical University Second Hospital (Other); The Third Affiliated Hospital of Beijing University (Unknown); Jiangsu Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Yinghao Sun, Professor, Changhai Hospital
Other Study IDs: POINT-2017
Record Dates: First submitted 2017-12-14; First posted 2018-01-09 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: male; lower urinary tract symptoms; comorbidities; chronic kidney diseases; urodynamics; medical therapy; surgical treatment
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood and urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oral medication group: Patients in this group will receive oral medications to treat lower urinary tract symptoms
  Interventions: Drug: Oral medications to treat lower urinary tract symptoms
- Surgical treatment group: Patients in this group receive minimal invasive transurethral prostate procedures.
  Interventions: Procedure: Minimal invasive transurethral prostate procedures

INTERVENTIONS:
Drug: Oral medications to treat lower urinary tract symptoms — Patients in this group will receive oral medication(s) depending on doctors' prescriptions.
  Groups: Oral medication group
Procedure: Minimal invasive transurethral prostate procedures — Patients in this group will receive surgical treatment.
  Groups: Surgical treatment group

SUMMARY:
The present is a multicenter, observational study organized by the Prostatic Obstruction Investigation Team (POInT), with a main purpose of looking into the current status and symptom progression of male lower urinary tract symptoms patients in China.

DETAILED DESCRIPTION:
Lower urinary tract symptoms (LUTS) is a common medical condition negatively affecting people's quality of life worldwide. LUTS may be caused by structural or functional abnormalities in 1 or more parts of the lower urinary tract, including bladder, prostate, internal and external urethral sphincter and distal urethra. Furthermore, evidence exists to demonstrate that LUTS is associate with lifestyle factors, systemic comorbidities and geriatric diseases, such as smoking, obesity, metabolic syndrome, chronic kidney diseases and chronic obstructive pulmonary disease etc. So far, there is lack of evidence to illustrate the symptom features and comorbidities among Chinese male LUTS patients. Therefore, this multicenter clinical study aims to investigate the present status and symptom progression among male LUTS patients in China.

ELIGIBILITY:
Inclusion Criteria:

1. Male, 45 years or older.
2. The presence of lower urinary tract symptoms, i.e. frequency, urgency, urge incontinence, dysuria, post-micturition dribble, etc.
3. All participants have signed the informed consent form.
4. Clinical data comes from 23 selected hospitals spread across China.

Exclusion Criteria:

1. Lower urinary tract symptoms as a result of urethral stricture, stone diseases, chronic prostatitis, space-occupying lesions etc.
2. Diagnosis or suspicion of renal, ureteral, bladder, prostate, urethral or pelvic tumor.
3. Known neurogenic or congenital lower urinary tract dysfunction.
4. Known urinary tract, prostate or pelvic surgical history.
5. Existence of anatomical abnormalities of the urinary tract (e.g. diverticulum of the bladder or urethra, ectopic ureteral orifice etc.).
6. The presence of acute conditions, such as, urinary tract infection, fever, heart failure etc.
7. Patients with poor compliance or cognitive competence.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese male, 45 year or elder, presenting lower urinary tract symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 11500 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
The changes of IPSS scores between baseline and follow-up | Measured at baseline and 6, 12, 18, 24, 36 months if oral medication is provided, or 1, 6, 18, 24 months after surgery.
  Measured using standard IPSS scoring system
The changes of nocturia symptoms between baseline and follow-up | Measured at baseline and 6, 12, 18, 24, 36 months if oral medication is provided, or 1, 6, 18, 24 months after surgery
  Measured using standard ICIQ-N-QoL score
The changes of erectile function between baseline and follow-up | Measured at baseline and 6, 12, 18, 24, 36 months if oral medication is provided, or 1, 6, 18, 24 months after surgery
  Measured using standard IIEF score
The changes of maximum flow rate (ml/s) between baseline and follow-up | Measured at baseline and 6, 12, 18, 24, 36 months if oral medication is provided or 1, 6, 18, 24 months after surgery
  Maximum flow rate will be measured using urinary flow study
The changes of post void residual volume (ml) between baseline and follow-up | Measured at baseline and 6, 12, 18, 24, 36 months if oral medication is provided or 1, 6, 18, 24 months after surgery
  post void residual volume (ml) will be measured using urinary flow study
The changes of detrusor pressure at maximum flow rate (cmH2O) between baseline and follow-up | Measured at baseline (if surgical treatment is required) and 1, 6, 18, 24 months after surgery
  It will be measured using pressure-flow study
The changes of prostate volume (ml) between baseline and follow-up | Measured at baseline and 6, 12, 18, 24, 36 months after oral medication treatment
  Prostate volume (ml) will be measured using transrectal prostate ultrasound and calculated as: prostate volume (ml) = length (mm) * width (mm) * height (mm) * 0.52
The changes of intravesical prostate protrusion (mm) between baseline and follow-up | Measured at baseline and 6, 12, 18, 24, 36 months after oral medication treatment
  Intravesical prostate protrusion (mm) will be measured using transrectal prostate ultrasound and calculated as the distance between the tip of the prostate median lobe and bladder neck

SECONDARY OUTCOMES:
The changes of Blood pressure between baseline and follow-up | Measured at baseline and 6, 12, 18, 24, 36 months if oral medication is provided or 1, 6, 18, 24 months after surgery.
  systolic pressure/ diastolic pressure in mmHg.
The changes of Blood lipid between baseline and follow-up | Measured at baseline and 6, 12, 18, 24, 36 months if oral medication is provided or 1, 6, 18, 24 months after surgery.
  The blood lipid level will be assessed using multiple serum parameters, namely, cholesterol (mmol/L), triglyceride (mmol/L), high-density lipoprotein (mmol/L), low-density lipoprotein (mmol/L), lipoprotein-a (mmol/L)
The changes of Blood glucose between baseline and follow-up | Measured at baseline and 6, 12, 18, 24, 36 months if oral medication is provided or 1, 6, 18, 24 months after surgery.
  The blood glucose level will be assessed using multiple serum parameters, namely, fast blood-glucose (mmol/L), glycosylated hemoglobin (%), glycated albumin (%)
The changes of Kidney function between baseline and follow-up | Measured at baseline and 6, 12, 18, 24, 36 months if oral medication is provided or 1, 6, 18, 24 months after surgery.
  The kidney function will be assessed using multiple serum and urine parameters, namely, serum creatinine (μmoI/L), cystatin-C (mg/L), eGRF (calculated via both CKD-EPI equation and MDRD equation), BUN (mmol/L), uric acid (μmoI/L), β2-MG (mg/L), NAG (U/L), Na (mmol/L), K (mmol/L), the degree of urine protein
The changes of PSA (ng/ml) between baseline and follow-up | Measured at baseline and 6, 12, 18, 24, 36 months if oral medication is provided or 1, 6, 18, 24 months after surgery.
  Serum PSA level will be measured to rule out prostate cancer
The changes of RBC (/HP) between baseline and follow-up | Measured at baseline and 6, 12, 18, 24, 36 months if oral medication is provided or 1, 6, 18, 24 months after surgery.
  Urine RBC will be measured to detect the incidence of urinary tract infection or tumor
The changes of WBC (/HP) between baseline and follow-up | Measured at baseline and 6, 12, 18, 24, 36 months if oral medication is provided or 1, 6, 18, 24 months after surgery.
  Urine WBC will be measured to detect the incidence of urinary tract infection

CONTACTS AND LOCATIONS:
Overall Officials: Yinghao Sun, MD, PhD, Study Chair — Changhai Hospital; Wei Xue, MD, PhD, Principal Investigator — RenJi Hospital; Qi-Xiang Song, MD,PhD, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Song QX, Zhang Y, Ye X, Xue W, Xu C, Xu J, Abrams P, Sun Y; Prostatic Obstruction Investigation Team (POInT). Current status and progression of lower urinary tract symptoms in Chinese male patients: the protocol and rationale for a nationwide, hospital-based, prospective, multicentre study. BMJ Open. 2019 Sep 27;9(9):e028378. doi: 10.1136/bmjopen-2018-028378. PMID 31562145

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-19): https://cdn.clinicaltrials.gov/large-docs/51/NCT03394651/Prot_SAP_000.pdf